CLINICAL TRIAL: NCT01767467
Title: Study to Evaluate Safety and Immunogenicity of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults Aged 18 Years and Older With Haematologic Malignancies
Brief Title: Study to Assess the Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine in Adults Aged 18 Years and Older With Blood Cancers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116428; 2012-003438-18 (EudraCT Number)
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Herpes Zoster
Keywords: Immunogenicity; Safety; Herpes zoster; Vaccination; Haematologic malignancies
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Vaccine Group (Experimental): Subjects will receive the candidate HZ vaccine (GSK 1437173A).
  Interventions: Biological: Herpes zoster vaccine (GSK 1437173A)
- Placebo Group (Placebo Comparator): Subjects will receive the placebo vaccine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Herpes zoster vaccine (GSK 1437173A) — 2 doses administered intramuscularly (IM) in deltoid region of non-dominant arm. Dose 1 administered at Day 0. Dose 2 administered 1-2 months post Dose 1.
  Arms: Vaccine Group
Drug: Placebo — 2 doses administered intramuscularly (IM) in deltoid region of non-dominant arm. Dose 1 administered at Day 0. Dose 2 administered 1-2 months post Dose 1.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of GSK Biologicals' vaccine GSK1437173A in subjects aged 18 years and older with blood cancers. The study will evaluate safety-related events and antibody and cellular immune responses to the study vaccine, as compared to placebo.

DETAILED DESCRIPTION:
Amendment to protocol posting:

Increase in sample size, update of country/region-specific information (Sections 5, 6 and 9).

Promotion of secondary to primary objective; related update of primary and secondary outcome measures (Sections 4 and 7).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male or female, aged 18 years or older at the time of study entry.
* Subject who has been diagnosed with one or more haematologic malignancies prior to the first vaccination and who is receiving, is scheduled to receive or has just finished immunosuppressive cancer therapy to treat this condition.
* Life expectancy greater than or equal to 12 months, as assessed by the investigator.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled inthe study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Subject diagnosed with chronic lymphocytic leukaemia (CLL) who is receiving only oral cancer therapy (subject receiving intra-venous cancer therapy for CLL or intra-venous cancer therapy in combination with oral therapy may be enrolled).
* Subject receiving radiotherapy alone as treatment for his/her haematologic malignancy.
* Planned haematopoietic stem cell transplant (HCT) during the study period. (If a HCT occurred prior to enrolment in the study, the subject may not receive study vaccine until at least 50 days after the transplant procedure).
* Human immunodeficiency virus (HIV) infection by clinical history.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period. However, the investigational use of a registered product to treat the subject's underlying disease, is allowed.
* Previous vaccination against HZ or varicella within the 12 months preceding the first dose of study vaccine/placebo.
* Planned administration during the study of a HZ or varicella vaccine (including an investigational or non-registered vaccine) other than the study vaccine.
* Occurrence of a varicella or HZ episode by clinical history within the 12 months preceding the first dose of study vaccine/placebo.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine.
* Administration or planned administration of a non-replicating vaccine within 8 days prior to or within 14 days after either dose of study vaccine.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions before Month 3 (i.e., 2 months after the last dose of study vaccine/placebo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2013-03-01; Primary Completion 2016-01-07 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (8):
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (4):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Coburg, Victoria
  - GSK Investigational Site, Wodonga, Victoria
- Belgium (6):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Jette
  - GSK Investigational Site, Leuven
- Canada (4):
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
- GSK Investigational Site, Prague, Czechia
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
- France (6):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Périgueux
  - GSK Investigational Site, Rouen
- GSK Investigational Site, Hong Kong, Hong Kong
- Italy (3):
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Novara, Piedmont
- New Zealand (2):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
- Pakistan (2):
  - GSK Investigational Site, Lahore
  - GSK Investigational Site, Multan
- GSK Investigational Site, Panama City, Panama
- Poland (3):
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Opole
  - GSK Investigational Site, Słupsk
- Russia (5):
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Singapore, Singapore
- South Korea (7):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jellanamdo
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Kyunggi-do
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Móstoles, Madrid
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Santander
- Sweden (4):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Uppsala
- Taiwan (4):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien
- GSK Investigational Site, Ankara, Turkey (Türkiye)
- United Kingdom (6):
  - GSK Investigational Site, Orpington, Kent
  - GSK Investigational Site, Airdrie, Lanarkshire
  - GSK Investigational Site, Swindon, Wiltshire
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Headington, Oxford
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505
- [Derived] Dagnew AF, Ilhan O, Lee WS, Woszczyk D, Kwak JY, Bowcock S, Sohn SK, Rodriguez Macias G, Chiou TJ, Quiel D, Aoun M, Navarro Matilla MB, de la Serna J, Milliken S, Murphy J, McNeil SA, Salaun B, Di Paolo E, Campora L, Lopez-Fauqued M, El Idrissi M, Schuind A, Heineman TC, Van den Steen P, Oostvogels L; Zoster-039 study group. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine in adults with haematological malignancies: a phase 3, randomised, clinical trial and post-hoc efficacy analysis. Lancet Infect Dis. 2019 Sep;19(9):988-1000. doi: 10.1016/S1473-3099(19)30163-X. Epub 2019 Aug 6. PMID 31399377

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 568 subjects enrolled, only 562 subjects received vaccination as per protocol and hence started the study.
Groups:
- GSK1437173A Group: Subjects who received GSK1437173A vaccine according to a 0, 1 Months schedule (The second dose of study vaccine could be administered 1 - 2 months after the first dose).
- Placebo Group: Subjects who received placebo doses according to a 0, 1 Months schedule (The second dose of placebo could be administered 1 - 2 months after the first dose).
Period: Vaccination Phase (up to Month 2)
Arm/Group | GSK1437173A Group | Placebo Group
Started | 283 | 279
Completed | 266 | 259
Not Completed | 17 | 20
Not completed — Adverse Event | 8 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 7 | 10
Not completed — Suspected Herpes Zoster episode | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Subject unavailable | 0 | 1
Period: End of Study Phase (up to Month 13)
Arm/Group | GSK1437173A Group | Placebo Group
Started | 283 | 279
Completed | 236 | 216
Not Completed | 47 | 63
Not completed — Adverse Event | 29 | 39
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 9 | 14
Not completed — Migrated/Moved from study area | 0 | 3
Not completed — Lost to Follow-up | 6 | 4
Not completed — Suspected Herpes Zoster episode | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Subject Unavailable | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Placebo Group | Total
Number analyzed (Participants) | 283 | 279 | 562
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (15.5) | 57.8 (14.9) | 57.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 114 | 228
  Male | 169 | 165 | 334
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage / African American | 1 | 1 | 2
  Geographic ancestry: American Indian or Alaskan Native | 0 | 1 | 1
  Geographic ancestry: Asian - Central / South Asian Heritage | 5 | 6 | 11
  Geographic ancestry: Asian - East Asian Heritage | 57 | 60 | 117
  Geographic ancestry: Asian - South East Asian Heritage | 4 | 1 | 5
  Geographic ancestry: White - Arabic / North African Heritage | 0 | 1 | 1
  Geographic ancestry: White - Caucasian / European Heritage | 198 | 186 | 384
  Geographic ancestry: Other | 7 | 12 | 19
  Geographic ancestry: Missing | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Response Rates (VRR) for Anti-glycoprotein E (Anti-gE) Antibody Concentrations
Description: Vaccine response rate refers to the percentage of subjects with a vaccine response, as determined by Enzyme-Linked Immunosorbent Assay (ELISA). Vaccine response was defined as: For initially seronegative subjects, antibody concentration at Month 2 greater than or equal to (≥) 4 fold the cut-off for Anti-gE [4x97 milli-international units per milliliter (mIU/mL)]. For initially seropositive subjects, antibody concentration at Month 2 ≥ 4 fold the pre-vaccination antibody concentration.
  This analysis was performed on subjects with haematologic malignancies excluding subjects with Non-Hodgkin B-cell Lymphoma and Chronic Lymphocytic Leukaemia.
Time Frame: At Month 2
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for Humoral immunogenicity, which included all subjects who met all eligibility criteria, who received the full vaccination course, complied with the protocol and and for whom data concerning immunogenicity outcome measures were available up to the Month 2 visit.
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- Placebo Group: Subjects who received placebo doses according to a 0, 1 Months schedule. (The second dose of placebo could be administered 1 - 2 months after the first dose).
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 148 | 130
Percentage | 80.4 [73.1 to 86.5] | 0.8 [0.0 to 4.2]

2. Primary Outcome: Adjusted Geometric Mean Concentration of Anti-gE Antibodies
Description: The Adjusted geometric mean concentration was measured in all subjects excluding those with Non-Hodgkin B-cell Lymphoma and Chronic Lymphocytic Leukaemia.
Time Frame: At Month 2
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for Humoral immunogenicity, which included all subjects who met all eligibility criteria, who received the full vaccination course, complied with the protocol and for whom data concerning immunogenicity outcome measures were available up to the Month 2 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 148 | 130
mIU/mL | 22132.9 [16642.8 to 32153.9] | 777.6 [702.8 to 860.3]
Statistical Analysis 1: Comparison: GSK1437173A Group vs Placebo Group; The objective aimed to evaluate anti-gE humoral immune responses at Month 2 following a two-dose administration of the GSK1437173A vaccine, as compared to placebo, in subjects with haematologic malignancies excluding subjects with Non-Hodgkin B-cell Lymphoma and Chronic Lymphocytic Leukaemia; Test type: Non-Inferiority — The objective was met if the lower limit of the 95% CI of the Geometric Mean (GM) ratio (GSK1437173A vaccine over placebo) for anti-gE ELISA antibody concentrations at Month 2 was greater than (>) 3; p < 0.0001, Repeated measurement model — The p-value is relative to the null hypothesis Ho: Vaccine / Placebo = 1; Adjusted Geometric Mean Concentration = 29.75, 95% CI 2-sided [21.09 to 41.96]

3. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine dose administered, who had their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 278 | 274
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 278 | 271
  Any Pain, Dose 1 | 199 | 26
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 Pain, Dose 1 | 16 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 278 | 271
  Any Redness, Dose 1 | 80 | 1
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 Redness, Dose 1 | 2 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 278 | 271
  Any Swelling, Dose 1 | 47 | 2
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 Swelling, Dose 1 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 255 | 248
  Any Pain, Dose 2 | 172 | 31
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 255 | 248
  Grade 3 Pain, Dose 2 | 20 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 255 | 248
  Any Redness, Dose 2 | 82 | 5
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 255 | 248
  Grade 3 Redness, Dose 2 | 10 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 255 | 248
  Any Swelling, Dose 2 | 42 | 1
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 255 | 248
  Grade 3 Swelling, Dose 2 | 5 | 0
  Any Pain, Across doses | 221 | 45
  Grade 3 Pain, Across doses | 29 | 0
  Any Redness, Across doses | 115 | 5
  Grade 3 Redness, Across doses | 12 | 0
  Any Swelling, Across doses | 63 | 2
  Grade 3 Swelling, Across doses | 5 | 0

4. Primary Outcome: Number of Days With Solicited Local Symptoms
Description: Solicited local symptoms: pain, redness, swelling and their number of days were recorded after each vaccination dose.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 278 | 271
Days
  Pain, Dose 1 | 3.0 [2.0 to 4.0] | 1.0 [1.0 to 2.0]
  Pain, Dose 2: number analyzed (Participants) | 255 | 248
  Pain, Dose 2 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Redness, Dose 1 | 3.0 [2.0 to 5.0] | 1.0 [1.0 to 1.0]
  Redness, Dose 2: number analyzed (Participants) | 255 | 248
  Redness, Dose 2 | 3.0 [2.0 to 5.0] | 4.0 [2.0 to 6.0]
  Swelling, Dose 1 | 3.0 [2.0 to 4.0] | 1.5 [1.0 to 2.0]
  Swelling, Dose 2: number analyzed (Participants) | 255 | 248
  Swelling, Dose 2 | 3.0 [2.0 to 4.0] | 4.0 [4.0 to 4.0]

5. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (included nausea, vomiting, diarrhoea and/or abdominal pain), headache, myalgia, shivering and fever [defined as oral, axillary or tympanic route measured temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 278 | 274
Participants
  Any fatigue, Dose 1: number analyzed (Participants) | 278 | 271
  Any fatigue, Dose 1 | 122 | 73
  Grade 3 fatigue, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 fatigue, Dose 1 | 11 | 8
  Related fatigue, Dose 1: number analyzed (Participants) | 278 | 271
  Related fatigue, Dose 1 | 37 | 11
  Any gastrointestinal, Dose 1: number analyzed (Participants) | 278 | 271
  Any gastrointestinal, Dose 1 | 48 | 24
  Grade 3 gastrointestinal, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 gastrointestinal, Dose 1 | 5 | 2
  Related gastrointestinal, Dose 1: number analyzed (Participants) | 278 | 271
  Related gastrointestinal, Dose 1 | 13 | 1
  Any headache, Dose 1: number analyzed (Participants) | 278 | 271
  Any headache, Dose 1 | 70 | 40
  Grade 3 headache, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 headache, Dose 1 | 3 | 3
  Related headache, Dose 1: number analyzed (Participants) | 278 | 271
  Related headache, Dose 1 | 29 | 10
  Any myalgia, Dose 1: number analyzed (Participants) | 278 | 271
  Any myalgia, Dose 1 | 80 | 35
  Grade 3 myalgia, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 myalgia, Dose 1 | 11 | 0
  Related myalgia, Dose 1: number analyzed (Participants) | 278 | 271
  Related myalgia, Dose 1 | 33 | 10
  Any shivering, Dose 1: number analyzed (Participants) | 278 | 271
  Any shivering, Dose 1 | 39 | 16
  Grade 3 shivering, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 shivering, Dose 1 | 2 | 0
  Related shivering, Dose 1: number analyzed (Participants) | 278 | 271
  Related shivering, Dose 1 | 14 | 2
  Any temperature, Dose 1: number analyzed (Participants) | 278 | 271
  Any temperature, Dose 1 | 33 | 15
  Grade 3 temperature, Dose 1: number analyzed (Participants) | 278 | 271
  Grade 3 temperature, Dose 1 | 0 | 1
  Related temperature, Dose 1: number analyzed (Participants) | 278 | 271
  Related temperature, Dose 1 | 18 | 3
  Any fatigue, Dose 2: number analyzed (Participants) | 255 | 247
  Any fatigue, Dose 2 | 126 | 67
  Grade 3 fatigue, Dose 2: number analyzed (Participants) | 255 | 247
  Grade 3 fatigue, Dose 2 | 16 | 6
  Related fatigue, Dose 2: number analyzed (Participants) | 255 | 247
  Related fatigue, Dose 2 | 49 | 13
  Any gastrointestinal, Dose 2: number analyzed (Participants) | 255 | 247
  Any gastrointestinal, Dose 2 | 53 | 16
  Grade 3 gastrointestinal, Dose 2: number analyzed (Participants) | 255 | 247
  Grade 3 gastrointestinal, Dose 2 | 5 | 2
  Related gastrointestinal, Dose 2: number analyzed (Participants) | 255 | 247
  Related gastrointestinal, Dose 2 | 20 | 4
  Any headache, Dose 2: number analyzed (Participants) | 255 | 247
  Any headache, Dose 2 | 90 | 42
  Grade 3 headache, Dose 2: number analyzed (Participants) | 255 | 247
  Grade 3 headache, Dose 2 | 10 | 3
  Related headache, Dose 2: number analyzed (Participants) | 255 | 247
  Related headache, Dose 2 | 42 | 9
  Any myalgia, Dose 2: number analyzed (Participants) | 255 | 247
  Any myalgia, Dose 2 | 93 | 25
  Grade 3 myalgia, Dose 2: number analyzed (Participants) | 255 | 247
  Grade 3 myalgia, Dose 2 | 14 | 5
  Related myalgia, Dose 2: number analyzed (Participants) | 255 | 247
  Related myalgia, Dose 2 | 50 | 7
  Any shivering, Dose 2: number analyzed (Participants) | 255 | 247
  Any shivering, Dose 2 | 48 | 7
  Grade 3 shivering, Dose 2: number analyzed (Participants) | 255 | 247
  Grade 3 shivering, Dose 2 | 9 | 0
  Related shivering, Dose 2: number analyzed (Participants) | 255 | 247
  Related shivering, Dose 2 | 27 | 1
  Any temperature, Dose 2: number analyzed (Participants) | 255 | 247
  Any temperature, Dose 2 | 51 | 11
  Grade 3 teamperature, Dose 2: number analyzed (Participants) | 255 | 247
  Grade 3 teamperature, Dose 2 | 3 | 0
  Related temperature, Dose 2: number analyzed (Participants) | 255 | 247
  Related temperature, Dose 2 | 28 | 3
  Any fatigue, Across doses | 162 | 102
  Grade 3 fatigue, Across doses | 23 | 10
  Related fatigue, Across doses | 63 | 22
  Any gastrointestinal, Across doses | 76 | 29
  Grade 3 gastrointestinal, Across doses | 9 | 3
  Related gastrointestinal, Across doses | 28 | 5
  Any headache, Across doses | 115 | 64
  Grade 3 headache, Across doses | 12 | 6
  Related headache, Across doses | 52 | 16
  Any myalgia, Across doses | 122 | 48
  Grade 3 myalgia, Across doses | 22 | 5
  Related myalgia, Across doses | 63 | 15
  Any shivering, Across doses | 69 | 18
  Grade 3 shivering, Across doses | 11 | 0
  Related shivering, Across doses | 36 | 2
  Any temperature, Across doses | 68 | 21
  Grade 3 temperature, Across doses | 3 | 1
  Related teamperature, Across doses | 36 | 4

6. Primary Outcome: Number of Days With Solicited General Symptoms
Description: Solicited general symptoms: fatigue, gastrointestinal symptoms, headache, myalgia, shivering, temperature and their number of days were recorded after each vaccination dose.
Time Frame: Withing the 7-day (Day 0-6) post-vaccination period
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 278 | 271
Days
  Fatigue, Dose 1 | 3.0 [1.0 to 6.0] | 3.0 [2.0 to 7.0]
  Fatigue, Dose 2: number analyzed (Participants) | 255 | 247
  Fatigue, Dose 2 | 3.0 [2.0 to 5.0] | 3.0 [1.0 to 7.0]
  Gastrointestinal symptoms, Dose 1 | 2.5 [1.0 to 5.0] | 3.5 [1.5 to 6.0]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 255 | 247
  Gastrointestinal symptoms, Dose 2 | 2.0 [1.0 to 3.0] | 6.0 [2.5 to 7.0]
  Headache, Dose 1 | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0]
  Headache, Dose 2: number analyzed (Participants) | 255 | 247
  Headache, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Myalgia, Dose 1 | 3.5 [2.0 to 5.5] | 3.0 [1.0 to 4.0]
  Myalgia, Dose 2: number analyzed (Participants) | 255 | 247
  Myalgia, Dose 2 | 2.0 [2.0 to 4.0] | 3.0 [1.0 to 7.0]
  Shivering, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.5]
  Shivering, Dose 2: number analyzed (Participants) | 255 | 247
  Shivering, Dose 2 | 1.0 [1.0 to 2.0] | 4.0 [2.0 to 4.0]
  Temperature, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Temperature, Dose 2: number analyzed (Participants) | 255 | 247
  Temperature, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0]

7. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study. It also included any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all all subjects with at least one vaccine dose administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 283 | 279
Participants
  Any AEs | 134 | 128
  Grade 3 AEs | 25 | 28
  Related AEs | 19 | 5

8. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A Serious adverse event (SAE) is any untoward medical occurrence that result in death, is life threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject. Related = SAEs assessed by the investigator as causally related to the study vaccination
Time Frame: From first vaccination up to 30 days post last vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine dose administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 283 | 279
Participants
  At least one SAE | 17 | 29
  Related SAEs | 0 | 0

9. Primary Outcome: Number of Subjects Reporting Any and Related Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Related = pIMds assessed by the investigator as causally related to the study vaccination
Time Frame: From first vaccination up to 30 days post last vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 283 | 279
Participants
  Any pIMDs | 1 | 0
  Related pIMDs | 0 | 0

10. Secondary Outcome: Vaccine Response Rate (VRR) for Anti-gE Antibody Concentrations
Description: Vaccine response rate refers to the percentage of subjects with a vaccine response, as determined by ELISA. Vaccine response was defined as: For initially seronegative subjects, antibody concentration at Month 2 ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/mL). For initially seropositive subjects, antibody concentration at Month 2 ≥ 4 fold the pre -vaccination antibody concentration. This analysis was performed on subjects with haematologic malignancies, excluding subjects with Non-Hodgkin B-cell Lymphoma.
Time Frame: At Month 2
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for Humoral immunogenicity, which included all subjects who met all eligibility criteria, received the full vaccination course, complied with the protocol and for whom data concerning immunogenicity outcome measures were available up to the Month 2 visit.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 184 | 165
Percentage | 69.0 [61.8 to 75.6] | 0.6 [0.0 to 3.3]

11. Secondary Outcome: Anti-gE Antibody Concentrations
Description: Antibody concentrations were determined by ELISA, presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL).This parameter was assessed in subjects with haematologic malignancies, excluding subjects with Non-Hodgkin B-cell Lymphoma.
Time Frame: At Month 2
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 184 | 165
mIU/mL | 15795.5 [11603.3 to 21502.2] | 791.6 [648.9 to 965.5]

12. Secondary Outcome: Time to Occurrence of Any Confirmed HZ Case
Description: Time to occurrence of any confirmed HZ case is expressed in terms of incidence rate of subjects with at least one event. Hence, person-year rate = number of episodes (n)/ sum of follow-up period (censored at the first occurrence of an event) expressed in years (T[year)]). Follow-up period starts Day 1 of vaccination.
  Any clinically suspected case of HZ (defined as (1) a new rash characteristic of HZ (e.g., unilateral, dermatomal and accompanied by pain broadly defined to include allodynia, pruritus or other sensations), or a vesicular rash suggestive of Varicella Zoster Virus (VZV) infection regardless of the distribution, and no alternative diagnosis; or (2) a clinical presentation (symptoms and/or signs) and specific laboratory findings suggestive of VZV infection in the absence of characteristic HZ or VZV rash.) The endpoint is confirmed in two ways: (1) By Polymerase Chain Reaction (PCR) or (2) By the HZ Ascertainment Committee. The PCR is used as primary classification method.
Time Frame: From Month 0 until study end (Month 13)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Person-year rate
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 283 | 279
Person-year rate | 0.020 [0.009 to 0.045] | 0.071 [0.045 to 0.111]

13. Secondary Outcome: Anti-gE Antibody Concentrations
Description: Antibody concentrations were determined by ELISA, presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). This parameter was assessed in all vaccinated subjects.
Time Frame: At Months 0, 1, 2 and 13
Population: The analysis was performed on the adapted ATP cohort for Humoral immunogenicity, which included all subjects who met all eligibility criteria, received the full vaccination course, complied with the protocol and for whom data concerning immunogenicity outcome measures were available up to the Month 13 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 217 | 198
mIU/mL
  Anti-gE, Month 0 | 964.0 [814.5 to 1140.8] | 883.7 [749.9 to 1041.4]
  Anti-gE, Month 1: number analyzed (Participants) | 215 | 196
  Anti-gE, Month 1 | 4216.5 [3328.6 to 5341.4] | 824.2 [699.4 to 971.3]
  Anti-gE, Month 2 | 13445.6 [10158.9 to 17795.6] | 832.0 [701.1 to 987.3]
  Anti-gE, Month 13: number analyzed (Participants) | 167 | 142
  Anti-gE, Month 13 | 5202.7 [4074.8 to 6642.8] | 895.4 [734.5 to 1091.5]

14. Secondary Outcome: Vaccine Response Rate (VRR) for Anti-gE Antibody Concentrations
Description: Vaccine response rate refers to the percentage of subjects with a vaccine response, as determined by ELISA. Vaccine response was defined as: For initially seronegative subjects, antibody concentration at Month 2 ≥ 4 fold the cut-off for anti-gE (4x97 mIU/mL). For initially seropositive subjects, antibody concentration at Month 2 ≥ 4 fold the pre -vaccination antibody concentration. Vaccine response was measured in all subjects.
Time Frame: At Months 1, 2 and 13
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 217 | 198
Percentage
  VRR, anti-gE, Month 1: number analyzed (Participants) | 215 | 196
  VRR, anti-gE, Month 1 | 44.2 [37.4 to 51.1] | 0.0 [0.0 to 1.9]
  VRR, anti-gE, Month 2 | 65.4 [58.7 to 71.7] | 0.5 [0.0 to 2.8]
  VRR, anti-gE, Month 13: number analyzed (Participants) | 165 | 140
  VRR, anti-gE, Month 13 | 52.1 [44.2 to 59.9] | 3.6 [1.2 to 8.1]

15. Secondary Outcome: Frequency of gE -Specific Cluster of Differentiation 4 (CD4) [2+] T-cells Expressing at Least 2 Activation Markers
Description: Among markers expressed were interferon-gamma (IFN-γ), interleukin-2 (IL-2), tumour necrosis factor-alpha (TNF-α) and cluster of differentiation 40 ligand (CD40L), as determined by in vitro intracellular cytokine staining (ICS).
Time Frame: At Months 0, 1, 2 and 13
Population: The analysis was performed on the adapted ATP cohort for Cell-Mediated Immunogenicity (CMI), which included all evaluable subjects included in the ATP cohort for Humoral immunogenicity analyses and included in the CMI sub-cohort.
Measure: Mean (Standard Deviation); unit: CD4 [2+] T-cells/million T-cells
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 58 | 51
CD4 [2+] T-cells/million T-cells
  CD4 [2+], Month 0: number analyzed (Participants) | 52 | 49
  CD4 [2+], Month 0 | 226.78 (659.84) | 147.30 (191.91)
  CD4 [2+], Month 1 | 1261.67 (2318.36) | 196.74 (332.52)
  CD4 [2+], Month 2: number analyzed (Participants) | 53 | 50
  CD4 [2+], Month 2 | 6083.98 (10467.57) | 318.20 (1000.90)
  CD4 [2+], Month 13: number analyzed (Participants) | 44 | 36
  CD4 [2+], Month 13 | 3626.87 (7758.18) | 181.23 (387.90)

16. Secondary Outcome: Vaccine Response Rates (VRR) for gE-specific CD4 [2+] T-cells, Expressing at Least 2 Activation Markers
Description: Among markers expressed were IFN-γ, IL-2, TNF-α and CD40L, as determined by in vitro ICS. Vaccine response was defined as:
  For initially subjects with pre-vaccination T-cell frequencies below the threshold, at least a 2-fold increase as compared to the threshold (2x<320> Events/106 CD4+ T cells).
  For initially subjects with pre-vaccination T-cell frequencies above the threshold, at least a 2-fold increase as compared to pre-vaccination T-cell frequencies.
Time Frame: At Months 1, 2 and 13
Population: The analysis was performed on the adapted ATP cohort for Cell Mediated Immunity (CMI), which included all evaluable subjects included in the ATP cohort for Humoral immunogenicity analyses and included in the CMI sub-cohort.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 48 | 47
Percentage
  CD4 [2+], Month 1 | 37.5 [24.0 to 52.6] | 2.1 [0.1 to 11.3]
  CD4 [2+], Month 2: number analyzed (Participants) | 43 | 44
  CD4 [2+], Month 2 | 83.7 [69.3 to 93.2] | 6.8 [1.4 to 18.7]
  CD4 [2+], Month 13: number analyzed (Participants) | 33 | 31
  CD4 [2+], Month 13 | 66.7 [48.2 to 82.0] | 6.5 [0.8 to 21.4]

17. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 8
Time Frame: From first vaccination at Month 0 up to study end at Month 13
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 283 | 279
Participants
  At least one SAE, up to Month 6 | 50 | 60
  Related SAEs, up to Month 6 | 0 | 1
  At least one SAE, up to Month 13 | 66 | 82
  Related SAEs, up to Month 13 | 1 | 1

18. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology
Time Frame: From first vaccination at Month 0 up to study end at Month 13
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 283 | 279
Participants
  Up to Month 6 | 3 | 1
  Up to Month 13 | 3 | 2

19. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-gE Antibodies
Description: GMCs of anti-gE antibodies were tabulated per study group and HZ confirmed/non-confirmed status and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Months 0 and 2
Population: This analysis was performed on the Cohort for correlate of protection, which included subjects from the Total vaccinated cohort receiving 2 vaccine doses and having no confirmed HZ-case before the Month 2 blood sampling.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Groups:
- GSK1437173A HZ Cases Sub-Group: Subjects who received GSK1437173A vaccine according to a 0, 1 Months schedule (The second dose of study vaccine could be administered 1 - 2 months after the first dose), with confirmed Herpes Zoster (HZ).
- GSK1437173A Non-HZ Cases Sub-Group: Subjects who received GSK1437173A vaccine according to a 0, 1 Months schedule (The second dose of study vaccine could be administered 1 - 2 months after the first dose), with non-confirmed Herpes Zoster (HZ).
- Placebo HZ Cases Sub-Group: Subjects who received placebo doses according to a 0, 1 Months schedule (The second dose of placebo could be administered 1 - 2 months after the first dose), with confirmed Herpes Zoster (HZ).
- Placebo Non-HZ Cases Sub-Group: Subjects who received placebo doses according to a 0, 1 Months schedule (The second dose of placebo could be administered 1 - 2 months after the first dose), with non-confirmed Herpes Zoster (HZ).
Arm/Group | GSK1437173A HZ Cases Sub-Group | GSK1437173A Non-HZ Cases Sub-Group | Placebo HZ Cases Sub-Group | Placebo Non-HZ Cases Sub-Group
Number analyzed (Participants) | 2 | 257 | 12 | 240
mIU/ml
  PRE | 115.9 [0.0 to 7406196] | 973.6 [835.6 to 1134.4] | 984.5 [500.7 to 1935.7] | 866.3 [745.5 to 1006.6]
  Month 2 | 184.0 [0.0 to 4187800000] | 12517.4 [9662.0 to 16216.6] | 960.5 [454.2 to 2031.1] | 802.9 [686.7 to 938.9]

20. Secondary Outcome: Mean Geometric Increase (MGI) of Anti-gE Antibody ELISA Concentrations
Description: MGI was tabulated per study group and HZ confirmed/non-confirmed status. MGI was defined as the Geometric mean of the within subject ratios of the post-vaccination reciprocal anti-gE concentration to the Month 0 reciprocal anti-gE concentration.
Time Frame: At Month 2
Population: This analysis was performed on the Cohort for correlate of protection, which included subjects from the Total vaccinated cohort receiving 2 vaccine doses and having no confirmed HZ-case before the Month 2 blood sampling, only on the subjects with available results at Month 2.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK1437173A HZ Cases Sub-Group | GSK1437173A Non-HZ Cases Sub-Group | Placebo HZ Cases Sub-Group | Placebo Non-HZ Cases Sub-Group
Number analyzed (Participants) | 2 | 253 | 12 | 233
Ratio | 1.59 [0.00 to 565.45] | 13.07 [9.93 to 17.22] | 0.98 [0.80 to 1.19] | 0.94 [0.88 to 1.00]

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited symptoms: within the 30-day (Days 0-29) post-vaccination period; SAEs: up to study end, at Month 13.
Arm/Group | GSK1437173A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 29/283 | 37/279
Serious Adverse Events (participants affected / at risk) | 66/283 | 82/279
Other Adverse Events (participants affected / at risk) | 252/283 | 146/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=283) | Placebo Group (N=279)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (16) | 11 (16)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Ophthalmoplegia (Eye disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adhesion (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Death neonatal (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 3 (3)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis fulminant (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (2) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (3) | 0 (0)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Corynebacterium bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ecthyma (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Perichondritis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 11 (12) | 11 (12)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (3) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 6 (6)
Septic shock (Infections and infestations) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 3 (4) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 8 (8)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blastic plasmacytoid dendritic cell neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Precursor t-lymphoblastic lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Stem cell transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=283) | Placebo Group (N=279)
Gastrointestinal disorder (Gastrointestinal disorders) | 76 (101) | 29 (40)
Chills (General disorders) | 69 (89) | 19 (24)
Fatigue (General disorders) | 163 (250) | 102 (140)
Pain (General disorders) | 221 (372) | 46 (60)
Pyrexia (General disorders) | 74 (96) | 24 (30)
Swelling (General disorders) | 63 (89) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 123 (175) | 48 (60)
Headache (Nervous system disorders) | 115 (166) | 65 (86)
Erythema (Skin and subcutaneous tissue disorders) | 116 (165) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.